CLINICAL TRIAL: NCT07029542
Title: A Mobile App-Based, Prospective, Observational Study to Evaluate Disease Burden and Treatment Patterns in C3 Glomerulopathy (C3G) in the US
Brief Title: Home Reported Outcomes in C3G Study
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLNP023B1US01
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: C3 Glomerulopathy
Keywords: Home reported outcomes (HRO),; NIS,; FACIT-F,; EQ-5D,; Symptoms,; Treatments

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- C3G: patients with confirmed diagnosis of C3 glomerulopathy (C3G)

SUMMARY:
The study aims to longitudinally capture the full spectrum of symptoms, treatment utilization, and overall Health-related Quality of Life (HRQoL) experienced by C3 glomerulopathy (C3G) patients and their caregivers. By primarily utilizing home reported outcomes (HRO) data on symptom burden and treatment usage, supplemented with patient-reported outcome (PRO) measures (collected at baseline and monthly), the study seeks to establish a new real-world data (RWD) source to understand symptom variability and HRQoL as reported by C3G patients and caregivers, including those taking iptacopan

DETAILED DESCRIPTION:
The study will be prospective and observational, conducted over an initial period of six months per individual from the point of study enrollment, with the potential option for participants to extend data collection beyond this period through reconsenting procedures. Participants will utilize the Folia mobile app to enroll, consent, and complete all study activities. A hybrid referral-based recruitment method will be used to identify eligible participants such as through the Novartis APPRISE and MPGN data platforms, clinician referrals, specialty pharmacy inserts, and community and advocacy groups. Participants will be asked to track routine treatment, symptoms, changes in treatment plans, and HRQoL using the Folia Health mobile app. Monthly survey check-ins will be conducted to capture additional data inputs such as patient-reported outcomes (PROs) data, which may be tokenized and integrated into the relevant Novartis APPRISE or MPGN data platform during and after their data collection period. Additional real-world evidence (RWE) datasets such as electronic health record (EHR), claims, or wearable/device data may also be linked to this prospective dataset. Data from integration sources would serve as a complement to the primary study dataset; integration does not affect study objectives or endpoints, which are achieved through HRO tracking data. Participants will be consented for tokenization and linkage through language built into the informed consent form.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will meet the following basic criteria:

* Clinical diagnosis of C3G, regardless of symptom, treatment, or transplant history
* Adult aged 18 or older; adult caregiver to an adult patient aged 18 or older; or adult caregiver to a pediatric patient under 18 years of age
* Able to provide informed consent
* Has access to technology (i.e. mobile phone, tablet) that facilitates their participation in the app-based study
* US-based with a proficient understanding of and ability to read the English language

The study team will aim to enroll and collect data on participants who are taking any form of treatment. Participants may be asked to recall the start date of taking their current therapy.

Diagnosis of C3G will be confirmed through self-reported screening procedures, patient-supplied documentation, and/or successful linkage of the patient's data with their record in a Novartis data platform. Confirmation of diagnosis for each participant will be reviewed by the Folia Health study team as part of standard validation procedures.

Exclusion Criteria:

Study participants who do not fit all inclusion criteria listed above are unable to participate in this study. Outside of the stated inclusion criteria, there is currently no other exclusion criteria in order to meet the exploratory nature of the primary endpoint. This includes treatment regimen; there is no exclusion criteria on the basis of treatment prescription or use.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample of 100 adults, caregivers of adults, or caregivers of children diagnosed with C3G across an initial 8-month enrollment period. The study team will aim to enroll approximately 50 participants who report taking iptacopan and 50 participants who are not taking a primary therapy of interest.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting the top 10 symptoms most frequently self-reported | 6 months
  Identification of the top 10 symptoms most frequently self-reported by participants, as well as the total number of participants reporting each of those symptoms
Participant average of self-reported severity of each of the top 10 symptoms | 6 months
  Across-participant average (and standard deviation) of self-reported severity of each of the top 10 symptoms over the course of the 6-month study
Within-participant variability in self-reported severity of each of the top 10 symptoms | 6 months
  Within-participant variability in self-reported severity of each of the top 10 symptoms over the course of the 6-month study

SECONDARY OUTCOMES:
Average temporal frequency of treatment administration | 6 months
  Average temporal frequency of treatment administration, for each primary treatment
Counts of patient-reported reasons for skipping treatment | 6 moths
  Identification and counts of patient-reported reasons for skipping treatment
Proportion of participants who report symptom burden | 6 months
  Differences in symptom burden for participants in each treatment group, including symptom occurrence (proportion of participants who report it), severity (when reported), and frequency (when reported).
Change in average symptom burden from pre-switch to post-switch, for participants who switched onto iptacopan during the study period | 6 months
  Change in average symptom burden (including occurrence, severity, and frequency) from pre-switch to post-switch, for participants who switched onto iptacopan during the study period, if there are enough participants who switch
Differences in number of participants by flare burden | 6 months
  Differences in number of participants in each treatment group who are classified as having a high vs moderate vs low flare burden
Change over time in monthly check-in responses assessing HRQoL | 6 months
  Change over time in monthly check-in responses assessing HRQoL, for participants in each treatment group (and in the transplant vs no transplant groups, if possible)
Differences in PRO scores | 6 months
  Differences in PRO scores, for participants in each treatment group (and in the transplant vs no transplant groups, if possible)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No